CLINICAL TRIAL: NCT05714059
Title: Safety and Effectiveness Evaluation of the MiniMed™ 780G System Used in Combination With the DS5 CGM
Brief Title: Safety and Effectiveness of the MiniMed™ 780G System With DS5 CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP337
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MiniMed™ 780G system with DS5 (Experimental): Subjects with type 1 diabetes wearing the MiniMed™ 780G insulin pump in combination with the DS5 CGM.
  Interventions: Device: Insulin Pump with Continuous Glucose Monitoring

INTERVENTIONS:
Device: Insulin Pump with Continuous Glucose Monitoring — MiniMed™ 780G insulin pump in combination with the DS5 CGM

SUMMARY:
The purpose of this study is to confirm the safety and effectiveness of the MiniMed 780G insulin pump used in combination with the DS5 CGM in type 1 diabetes adult and pediatric subjects in a home setting.

DETAILED DESCRIPTION:
This study is a multi-center, single arm study in insulin-requiring adult and pediatric subjects with type 1 diabetes on the MiniMed 780G system using DS5 as well as Medtronic Extended infusion set and reservoir. The run-in period and study period will be approximately 120 days long.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 - 80 years at time of screening.
2. Has a clinical diagnosis of type 1 diabetes:

   1. 14 - 80 years of age: A clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
   2. 7 - 13 years of age: A clinical diagnosis of type 1 diabetes for 1 year or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Does not require a legally authorized representative to consent on their behalf due to mental or intellectual disability.
4. Subject or parent/caregiver is literate and able to read the language offered in the pump or pump materials.
5. Subject and/or legally authorized representative is willing to provide informed consent for participation.
6. Is willing to perform fingerstick blood glucose measurements as needed.
7. Is willing to wear the system continuously throughout the study.
8. Must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units.
9. Has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by Central Lab) at time of screening visit.
10. Has thyroid-stimulating hormone (TSH) in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
11. Uses pump therapy for greater than 6 months prior to screening (with or without CGM experience).
12. Is willing to upload data from the study pump, must have Internet access, and a computer system, or compatible smartphone that meets the requirements for uploading the study pump.
13. Is willing to take one of the following insulins and can financially support the use of insulin preparations as required by the study:

    1. Humalog (insulin lispro injection)
    2. NovoLog (insulin aspart injection)
    3. Admelog (insulin lispro injection)

Exclusion Criteria:

1. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   1. Medical assistance (i.e., Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma
   3. Seizures
2. Has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes.
3. Has had DKA in the last 6 months prior to screening visit.
4. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
5. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Is female of child-bearing potential and result of pregnancy test is positive at screening.
7. Is sexually active female of child-bearing potential and is not using a form of contraception deemed reliable by the investigator.
8. Is female and plans to become pregnant during the course of the study.
9. Is being treated for hyperthyroidism at time of screening.
10. Has diagnosis of adrenal insufficiency.
11. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
12. Is using hydroxyurea at time of screening or plans to use it during the study.
13. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
14. Has used a MiniMed 780G pump prior to screening.
15. Is currently abusing illicit drugs.
16. Is currently abusing marijuana.
17. Is currently abusing prescription drugs.
18. Is currently abusing alcohol.
19. Using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening.
20. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
21. Has elective surgery planned that requires general anesthesia during the course of the study.
22. Has sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
23. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
24. Is diagnosed with current eating disorder such as anorexia or bulimia.
25. Has been diagnosed with chronic kidney disease that results in chronic anemia.
26. Has a hematocrit that is below the normal reference range of lab used.
27. Is on dialysis.
28. Has serum creatinine of >2 mg/dL.
29. Has celiac disease that is not adequately treated as determined by the investigator.
30. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
31. Has had history of cardiovascular event 1 year or more from the time of screening without

    1. a normal EKG and stress test within 6 months prior to screening or during screening or
    2. clearance from a qualified physician prior to receiving the study devices if there is an abnormal EKG or stress test.
32. Has 3 or more cardiovascular risk factors listed below without a normal EKG within 6 months prior to screening or during screening or clearance from a qualified physician if there is an abnormal EKG:

    * Age >35 years
    * Type 1 diabetes of >15 years' duration
    * Presence of any additional risk factor for coronary artery disease
    * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
    * Presence of peripheral vascular disease
    * Presence of autonomic neuropathy
33. Is a member of the research staff involved with the study.
34. Is a Medtronic Diabetes employee or their immediate family member (excluding adult children and/or adult siblings).

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Medical Investigations, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - University of California San Francisco (UCSF) The Madison Clinic for Pediatric Diabetes, San Francisco, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of South Florida (USF) Diabetes Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Joslin Diabetes Center, Boston, Massachusetts
  - Park Nicollet International Diabetes Center, Saint Louis Park, Minnesota
  - Childrens Hospital and Clinics of Minnesota, Saint Paul, Minnesota
  - New York University (NYU) Langone Hospital Long Island, Mineola, New York
  - Northwell Health for Cohen Children's Medical Center of New York, New Hyde Park, New York
  - University Hospitals Rainbow Babies & Childrens Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - Seattle Childrens Hospital, Seattle, Washington
  - Multicare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 250 subjects (125 with age 7-17 and 125 with age 18-80) enrolled at the beginning, with 20 (7 with age7-17 and 13 with age 18-80) screen failure, 8 subjects (6 with age 7-17 and 2 with age 18-80) early withdrawn, 222 subjects (112 with age 7-17 and 110 with age 18-80) were left as the Intention to Treat Population and started the study.
Groups:
- Subjects 7-17 Years of Age: Subjects 7-17 years of age wearing MiniMed™ 780G System With DS5 CGM
- Subjects 18-80 Years of Age: Subjects 18-80 years of age wearing MiniMed™ 780G System With DS5 CGM
Period: Overall Study
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Started | 112 | 110
Completed | 107 | 105
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — WITHDRAWAL BY PARENT/GUARDIAN | 3 | 0
Not completed — TECHNICAL PROBLEMS | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.0) | 46.7 (15.8) | 29.8 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 56 | 104
  Male | 64 | 54 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 101 | 105 | 206
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 95 | 104 | 199
  More than one race | 8 | 1 | 9
  Unknown or Not Reported | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.9 (4.8) | 28.8 (5.9) | 25.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Change in HbA1c
Description: The overall mean change in HbA1c from baseline to end of 3-month study period. Non-inferiority test.
Time Frame: 3 months
Population: Intention to Treat Population" to "Intention to Treat Population and HbA1c at exit were collected. HbA1c at exit were collected from 217 subjects in intention to treat population (111 subjects with age 7-17 and 106 subjects with age 18-80)
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 111 | 106
percentage of HbA1c | -0.4 (0.8) | -0.7 (0.7)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c, from baseline to end of 3-month study period was estimated and compared by a non-inferiority test to the threshold of -0.38% with a margin of 0.4%; p < 0.001, Wilcoxon (Mann-Whitney); Mean difference from baseline to exit = -0.4, 95% CI 2-sided [-0.6 to -0.3] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c from baseline to end of 3-month study period was estimated and compared by a non-inferiority test to the threshold of -0.50% with a margin of 0.4%. A significance level of 0.025 (one-sided) was used; p < 0.001, t-test, 1 sided; Mean difference from baseline to exit = -0.7, 95% CI 2-sided [-0.8 to -0.6] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint

2. Primary Outcome: Primary Effectiveness Endpoint for Age 18-80 - Percent of Time in Range (TIR 70-180 mg/dL)
Description: Age 18-80: The mean % of time in range (TIR 70-180 mg/dL). Non-inferiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: Intention to Treat Population and Time in range metric were available from last 6-7 weeks of 3 month study period. Time in range metrics from last 6-7 weeks of 3 month study period were available from 216 subjects in intention to treat population (109 subjects with age 7-17 and 107 subjects with age 18-80)
Measure: Mean (Standard Deviation); unit: percentage of Time in Range (TIR 70-180)
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 109 | 107
percentage of Time in Range (TIR 70-180) | 71.4 (9.9) | 80.2 (8.1)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL) was estimated and compared by a non-inferiority test to the threshold of 65.3% with a margin of 7.5%; p < 0.001, Wilcoxon (Mann-Whitney); Mean value (Final Values) = 71.4, 95% CI 2-sided [69.5 to 73.3] — This is one arm study, the Percent of Time in Range (TIR 70-180 mg/dL) from the last 6-7 weeks of 3 month study period was summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL) was estimated and compared by a non-inferiority test to the threshold of 73.7% with a margin of 7.5%; p < 0.001, t-test, 1 sided; Mean value (Final Values) = 80.2, 95% CI 2-sided [78.7 to 81.8] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Secondary Effectiveness Endpoint 1 - Percent of Time in Hypoglycemia (< 54 mg/dL)
Description: The mean % of time in hypoglycemia (< 54 mg/dL) . Non-inferiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: Intention to Treat Population and Time in hypoglycemia metrics were available from last 6-7 weeks of 3 month study period. Time in hypoglycemia metrics from last 6-7 weeks of 3 month study period were available from 216 subjects in intention to treat population (109 subjects with age 7-17 and 107 subjects with age 18-80)
Measure: Mean (Standard Deviation); unit: percentage of Time in Hypoglycemia(< 54)
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 109 | 107
percentage of Time in Hypoglycemia(< 54) | 0.4 (0.3) | 0.2 (0.4)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % time in hypoglycemia (< 54 mg/dL) was estimated and compared by a non-inferiority test to the threshold of 0.71% with a margin of 2%; p < 0.001, Wilcoxon (Mann-Whitney); Mean value (Final Values) = 0.4, 95% CI 2-sided [0.3 to 0.4] — This is one arm study, the Percent of Time in Hypoglycemia (< 54 mg/dL) from last 6-7 weeks of 3 month study period was estimated for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % time in hypoglycemia (< 54 mg/dL) was estimated and compared by a non-inferiority test to the threshold of 0.86% with a margin of 2%; p < 0.001, Wilcoxon (Mann-Whitney); Mean value (Final Values) = 0.2, 95% CI 2-sided [0.1 to 0.3] — This is one arm study, the Percent of Time in Hypoglycemia (< 54 mg/dL) were summarized from last 6-7 weeks of 3 month study period for this endpoint

4. Secondary Outcome: Secondary Effectiveness Endpoint 2 - Percent of Time in Range (TIR 70-180 mg/dL)
Description: The mean % of time in range (TIR 70-180 mg/dL ).Superiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Time in Range (70-180)
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 109 | 107
percentage of Time in Range (70-180) | 71.4 (9.9) | 80.2 (8.1)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL) was estimated and compared to a threshold of 65.3% by a simple superiority test; p < 0.001, Wilcoxon (Mann-Whitney); Mean value (Final Values) = 71.4, 95% CI 2-sided [69.5 to 73.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL) was estimated and compared to a threshold of 73.7% by a simple superiority test; p < 0.001, t-test, 1 sided; Mean value (Final Values) = 80.2, 95% CI 2-sided [78.7 to 81.8] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 month Study period
Description: Only the adverse event in the study period are posted here.
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/112 | 3/110
Other Adverse Events (participants affected / at risk) | 46/112 | 35/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age (N=112) | Subjects 18-80 Years of Age (N=110)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age (N=112) | Subjects 18-80 Years of Age (N=110)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Illness (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Infusion site dermatitis (General disorders) | 1 (1) | 1 (1)
Infusion site haemorrhage (General disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 1 (1)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 2 (2) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Medical device site pruritus (General disorders) | 0 (0) | 1 (2)
Medical device site reaction (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (3) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal foot infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 4 (12) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Medical device site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Purulent discharge (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Vitamin B12 increased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dysphemia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to publish until 12 months from trial completion or until sponsor publishes multi-center results, whichever occurs first. In either case, sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period more than 60 days but less than or equal to 180 days from the date that the communication is submitted to sponsor for review. Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT05714059/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT05714059/SAP_001.pdf